CLINICAL TRIAL: NCT06116357
Title: The Safety and Efficacy of Carotid Body Modulation Therapy in Hypertensive Patients by External Ultrasonic Micro-bubble
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jing Huang (Other)
Collaborators: The Second Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Sponsor-Investigator, Jing Huang, Prof., The Second Affiliated Hospital of Chongqing Medical University
Organization: The Second Affiliated Hospital of Chongqing Medical University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-78
Record Dates: First submitted 2023-06-19; First posted 2023-11-03 (Actual); Last update posted 2023-11-03 (Actual); Status verified 2023-10

CONDITIONS: Primary Hypertension
Keywords: Carotid body modulation therapy; Hypertension; Carotid body activity; Carotid body volume; Ultrasonic micro-bubble
MeSH Terms: conditions — Essential Hypertension; Hypertension

STUDY DESIGN:
Intervention Model Description: primary hypertensive patients
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Health volunteers (Other): Evaluate the CB activity of health volunteers as the control
  Interventions: Device: External Ultrasonic Micro-bubble

INTERVENTIONS:
Device: External Ultrasonic Micro-bubble — The enrollmented hypertensive patients should aceepted CB modulation therapy by external ultrasonic micro-bubble

SUMMARY:
The investigators intend to find a noninvasive method for CB modulation therapy and find a simple and convenient indicator for assessing CB activity. This study was designed to evaluate the safety and efficacy of carotid body modulation therapy in hypertensive patients by external ultrasonic micro-bubble and also identify the association between CB volume and CB activity.

DETAILED DESCRIPTION:
Carotid body (CB) hyperactivity, with excessive afferent discharge signal to the respiratory centre anautonomic sympathetic nuclei, can result in hyperventilation and sympathetic hyperactivity. And previous studies have found that CB hyperactivity was common in several kinds of cardiovascular diseases and the investigators also found that CB was obviously enlargement in hypertension and other cardiovascular diseases. Hence, CB might play an important role in the development of these cardiovascular diseases. Moreover, Resection of CB or blockade of P2X3 receptors in CB significantly reduced blood pressure (BP) and muscle sympathetic nerve activity (MSNA) in patients with hypertension. Therefore, CB may be a promising therapeutic target for hypertension. However, the following questions about CB are needed to be addressed urgently. First, the CB volume enlargement may be a promising indicator for selection appropriate patients for CB modulation therapy, but its relationship with the CB hyperactivity is still unclear. Second, although CB resection could significantly reduce BP in hypertensive patients, but the invasive therapy and completely resection may result in severe adverse events.

Based on the aforementioned questions, to find a simple and convenient indicator for assessing CB activity and find a noninvasive method for CB modulation therapy, the investigators designed this study to identify the association between CB volume and CB activity in hypertensive patients and also evaluated the safety and efficacy of carotid body modulation therapy in hypertensive patients by external ultrasonic micro-bubble.

ELIGIBILITY:
Inclusion Criteria:

* Hypertensive patients for CB modulation therapy

  1. Two or more antihypertensive medications that had been prescribed at least 50% of the manufacturer's maximum dose for at least 2 consecutive weeks before study; Patients take an angiotensin-converting enzyme inhibitor (ACEI) (or angiotensin-ⅱ receptor antagonist (ARB)) and calcium channel blocker (CCB) (or thiazide diuretic) ; Office systolic blood pressure (SBP)≥150 mmHg and <180mmHg.

     2.24-hour ambulatory systolic blood pressure: ≥135 mmHg and <170 mmHg

  3.A history of primary hypertension was recorded. 4.Patients who can understand the purpose of the trial, voluntarily participate and sign informed consent, and are willing to cooperate with clinical follow-up
* Patients for CB Volume and activity evaluation Hypertension group

  1. Primary hypertension patients agrees to take part in this study and perform CB MRI, ultrasound, CB activity tests and sign the informed consent.
  2. The office blood pressure of patients ≥ 140/90 mmHg; the patents were diagnosed hypertension and are taking anti-hypertensive drugs could also include, although the office blood pressure < 140/90 mmHg.
  3. The CB could be detected by carotid ultrasound or MRI. Control group

  <!-- -->

  1. The volunteers agree to take part in this study and perform CB MRI, ultrasound, CB activity tests and sign the informed consent.
  2. The volunteers are healthy.

Exclusion Criteria:

* Hypertensive patients for CB modulation therapy

  1. Carotid body anatomy is not eligible for treatment: ultrasound examination before treatment fail to find carotid body at carotid artery bifurcation.
  2. Carotid body anatomical heterotopic is difficult to select or unsuitable for ultrasound irradiation.
  3. Carotid anatomy that does not meet treatment conditions: severe carotid stenosis or occlusion.
  4. Carotid ulcer.
  5. Severe tortuosity of carotid artery
  6. After carotid artery stenting or stripping
  7. Other conditions that are not suitable for carotid intervention
  8. Glomerular filtration rate (eGFR) <45 mL/min / 1.73 m2
  9. Have type 1 diabetes or poorly controlled type 2 diabetes (defined as plasma HbA1c≥ 9.0% or 24-hour urinary protein quantity >1g/24h or proliferative retinal lesions)
  10. postural hypotension.
  11. Recent vascular events: Experienced acute myocardial infarction, unstable angina, syncope, or cerebrovascular accident within 3 months of the screening period.
  12. Suspected secondary hypertension.
  13. Respiratory support: The individual requires long-term oxygen support or mechanical ventilation (except for nighttime breathing support only because of sleep apnea).
  14. Life expectancy <1 year.
  15. A woman who is pregnant, breastfeeding, or planning to become pregnant.
  16. Subjects who are currently enrolled in another clinical trial and have not completed the primary endpoint.
  17. Allergic to contrast media.
  18. The investigators judged the patients' poor compliance and other reasons for not being suitable for participants in the trial.
  19. Any other conditions that the investigator did not consider appropriate to participate in the trial.
* Patients for CB Volume and activity evaluation

  1. the CB could not be detected by carotid ultrasound or MRI.
  2. The patients have secondary hypertension, heart failure.
  3. The patients have type 1diabetes mellitus, CB tumor.
  4. The patients were diagnosed as OSAS.
  5. The patients have severe chronic constructive pulmonary disease, interstitial lung disease or other severe lung diseases.
  6. Women who are pregnant, breastfeeding, or planning to become pregnant.
  7. Patients with other conditions which are not appropriate for enrollment judged by the investigators.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
The change from baseline 24-hour mean ambulatory SBP at 6 months | 6 months
  The investigators would evaluate the change from baseline 24-hour mean ambulatory SBP at 6 months after CB modulation therapy.
The change from baseline daytime mean ambulatory SBP at 6 months | 6 months
  The investigators would evaluate the change from baseline daytime mean ambulatory SBP at 6 months after CB modulation therapy.
The control rate of hypertension at 6 month | 6 months
  The investigators would evaluate the control rate of hypertension at 6 month after CB modulation therapy.

SECONDARY OUTCOMES:
The change from baseline CB activity at 6months | 6 months
  The investigators would evaluate the change from baseline CB activity at 6months in hypertension patients after CB modulation therapy.
The change from baseline CB volume at 6months | 6 months
  The investigators would evaluate the change from baseline CB volume at 6months in hypertension patients after CB modulation therapy.
The change from baseline 24-hour mean ambulatory DBP at 6 months | 6 months
  The investigators would evaluate the change from baseline 24-hour mean ambulatory DBP at 6 months after CB modulation therapy.
The change from baselines office SBP and DBP at 6 months | 6 months
  The investigators would evaluate the change from baselines office SBP and DBP at 6 months after CB modulation therapy.
The incidence of CB modulation therapy associated adverse events including MACE events, hypotension, carotid artery stenosis and hyoxemia at 6 months | 6 months
  The investigators would evaluate the incidence of CB modulation therapy associated adverse events including MACE events, hypotension, carotid artery stenosis and hyoxemia at 6 months after CB modulation therapy.
The differences of CB volume between healthy volunteers and hypertension patients | at baseline
  The investigators would evaluate the differences of CB volume between healthy volunteers and hypertension patients at baselines.
The differences of CB activity between healthy volunteers and hypertension patients | at baseline
  The investigators would evaluate the differences of CB activity between healthy volunteers and hypertension patients at baselines.
The correlation analysis of heart rate variability and CB activity in hypertension patients at baseline | at baseline
  The investigators would evaluate the association between heart rate variability and CB activity in hypertension patients at baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Jing Huang, MD, Principal Investigator — The Second Affiliated Hospital of Chongqing Medcial University
Locations (1):
- The Second Affilated Hospital of Chongqing Medical Universty, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No
We may share the IPD when the study was completely finished.

REFERENCES:
- [Background] Xue Q, Wang R, Wang L, Xiong B, Li L, Qian J, Hao L, Wang Z, Liu D, Deng C, Rong S, Yao Y, Jiang Y, Zhu Q, Huang J. Downregulating the P2X3 receptor in the carotid body to reduce blood pressure via acoustic gene delivery in canines. Transl Res. 2021 Jan;227:30-41. doi: 10.1016/j.trsl.2020.06.005. Epub 2020 Jun 14. PMID 32554072
- [Background] Del Rio R, Marcus NJ, Schultz HD. Carotid chemoreceptor ablation improves survival in heart failure: rescuing autonomic control of cardiorespiratory function. J Am Coll Cardiol. 2013 Dec 24;62(25):2422-2430. doi: 10.1016/j.jacc.2013.07.079. Epub 2013 Sep 4. PMID 24013056
- [Background] Iturriaga R, Del Rio R, Idiaquez J, Somers VK. Carotid body chemoreceptors, sympathetic neural activation, and cardiometabolic disease. Biol Res. 2016 Feb 26;49:13. doi: 10.1186/s40659-016-0073-8. PMID 26920146
- [Background] Niewinski P, Janczak D, Rucinski A, Tubek S, Engelman ZJ, Piesiak P, Jazwiec P, Banasiak W, Fudim M, Sobotka PA, Javaheri S, Hart EC, Paton JF, Ponikowski P. Carotid body resection for sympathetic modulation in systolic heart failure: results from first-in-man study. Eur J Heart Fail. 2017 Mar;19(3):391-400. doi: 10.1002/ejhf.641. Epub 2016 Sep 20. PMID 27647775
- [Result] Tan J, Xiong B, Zhu Y, Yao Y, Qian J, Rong S, Yang G, Zhu Q, Jiang Y, Zhou Q, Liu D, Deng C, Ran H, Wang Z, He T, Huang J. Carotid body enlargement in hypertension and other comorbidities evaluated by ultrasonography. J Hypertens. 2019 Jul;37(7):1455-1462. doi: 10.1097/HJH.0000000000002068. PMID 30925145